### **Consent Form**

# Study Title:

Feasibility a combining rehabilitation program at field exercises and tele-exercises to enhance daily life activities to rural women in Iraq

# Purpose:

We prepared a combining rehabilitation program (CRP) incorporate and safe rehabilitative exercise at home with popular games at field that suit the rural women to improve their quality of life and support them physically. Also, we are studying whether a program of in-person field exercises and remote tele-exercises can improve daily life activities for rural women and reduce discomfort among rural women in Iraq.

#### What You Will Do:

Attend exercise sessions in your community and do home exercises via phone/WhatsApp. Complete simple tests before and after the program. Program lasts about [12] weeks. We obtained the ethical approval from the scientific research committee for Athletic Sciences Department of College of Physical Education and Sport Sciences at University of Mosul. Decision number: UoM.S-1/24 in Date: 02/June/2024.

#### Possible Risks:

Mild muscle soreness or tiredness. Rare risk of injury if exercises are not done as instructed.

### Possible Benefits:

- -Mild muscle soreness or fatigue may occur after exercise.
- -There is a small risk of injury if exercises are not done as instructed.
- -Some participants may experience inconvenience due to scheduling or travel for field sessions.

| Confidentiality: |
|---|
| Your name will not appear in reports. Your information will be kept private. |
| Voluntary: |
| Joining is your choice. You can stop at any time without penalty. |
| Contact: |
| Munib A FATHE |
| Assistant Prof. PhD. Injuries Rehabilitation and Therapeutic Sport University of Mosul, College of Physical Education and Sport Sciences, Mosul, Iraq Address: Avro-city, Dohuk, Kurdistan Region, IRAQ Tel: WhatsApp: +96407701680770 Email: m.a.fathi@uomosul.edu.iq |
| Consent: |
| I have read and understood the above information and agree to take part. |

Participant Name: \_\_\_\_\_\_ Date: \_\_\_\_\_

Researcher Name: \_\_\_\_\_ Date: \_\_\_\_\_

Signature: